CLINICAL TRIAL: NCT00294476
Title: A One Arm, Open Label,Multi - Center Phase II Study to Evaluate the Safety and Efficacy of IVIG in the Treatment of Various Metastatic Solid Tumors for Which There is no Better Alternate Treatment
Brief Title: IVIG in the Treatment of Metastatic Cancers of the Prostate, Colon and Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GammaCan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCan-01
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-09

CONDITIONS: Cancer of Colon; Malignant Melanoma; Urologic Cancer
Keywords: IVIg; Cancer; Melanoma
MeSH Terms: conditions — Colonic Neoplasms; Melanoma; Urologic Neoplasms; Neoplasms | interventions — Immunoglobulins, Intravenous; Biological Therapy

INTERVENTIONS:
Drug: IVIG
Procedure: Biological Therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IVIG in the treatment of metastatic cancer of the prostate, colon and melanoma.

DETAILED DESCRIPTION:
This study is a one arm, open label, multi-center, phase II study. Its aim is to evaluate the safety and efficacy of IVIG administered as treatment for metastasis solid tumors. IVIG was proven as affecting the growth of tumor metastasis in animals' models.

Study population is including male or female, 18 and older, diagnosed as having a primary tumor (colon, melanoma or prostate) with measurable metastasis (according to the RECIST criteria) in soft tissues and/ or tumor markers in prostate cancer, for which there is no better alternate treatment.

The patients receive the IVIG calculated as 1g/kg/bodyweight per cycle (defined as every 21 days) until progression disease is noted. All patients are being followed for a period of 6 months after patient's withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age.
* Histological confirmed diagnosis of a prostate adenocarcinoma, melanoma or colon cancer
* At least one measurable site of disease as evidenced by CT or MRI, RECIST criteria in soft tissue OR lymph nodes and OR tumor markers as appropriate
* Rising PSA in 3 consecutive weeks taken at least one week apart with a value of at least 5 ng/mL
* Testosterone that is less than 50 ng/dL in prostate patients
* Prostate cancer patients receiving radiation therapy that is less than 30% of pelvic/total bone mass and where acute radiation toxicity is resolved
* ECOG Performance status 0- 2
* WBC > 1,500 cells/mm3, hemoglobin > 9 g/dL, and platelets > 100,000 cells/mm3 and < 500,000 cells/mm3
* Adequate renal function: serum creatinine < 2.0 mg/dL, or CCT>= 50 ml/min
* Life expectancy of at least 3 months
* Willing to participate in a 6 month follow-up
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Post menopausal women must be amenorrheic for at least 12 months to be considered of non- childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Patients who have given written informed consent

Exclusion Criteria:

* Patients suffering from primary or metastatic brain or spinal tumor.
* Patients with known sensitivity to any of the components of the IVIG formulation excipients.
* IgA levels <=60mg/dl .
* Treatment with IVIG 6 months prior to study start
* Patients that are with known seropositivity for HIV or with a known diagnosis of human immunodeficiency virus (HIV) infection. (AIDS)
* Patients with significant diseases, active infection or uncontrolled medical condition (e.g., pulmonary, neurological, cardiovascular, gastrointestinal, genitourinary) considered high risk for investigational new drug treatment/ who in the opinion of the investigator would be excluded from the study
* Female patients who are pregnant or breast-feeding.
* Patient has a severe and/or uncontrolled renal failure.
* Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent and who in the opinion of investigator, are unlikely to comply with the study protocol
* Patients who are currently participating or have participated in another clinical trial in the last 30 days.
* Patients who have undergone chemotherapy in the last 4 weeks
* Patients who are being treated with antibiotic treatment for an active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07

PRIMARY OUTCOMES:
1. Tumor response is measured at baseline and evaluated every 3 treatment cycles (9 weeks) by RECIST(CT or MRI measurements), Time to Progression
and Serum tumor markers as appropriate CEA, PSA. Additionally, ECOG performance status is evaluated before each treatment cycle

SECONDARY OUTCOMES:
Secondary efficacy measurements: Overall survival, Karnofsky Performance Status is evaluated at baseline and before each treatment cycle and Quality of life questionnaires is completed and evaluated at baseline and every 3 treatment cycles (9 weeks)
Safety assessments include Adverse events and laboratory values which are measured and evaluated before every treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Dan Aderka, M.D., Principal Investigator — Oncology institute, Sheba Madical Center
Locations (3):
- Israel (3):
  - Ella Institute, Oncology institute, Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Oncology Institute, Sheba Medical Center, Tel Litwinsky, Ramat Gan
  - Oncology institute, Shaare Zedek Medical Center, Jerusalem